CLINICAL TRIAL: NCT04666129
Title: A Phase 1, Three-Part, Open-Label, Parallel-Cohort Safety and Tolerability Study of Relugolix in Combination With Abiraterone Acetate Plus a Corticosteroid, Apalutamide, or Docetaxel With or Without Prednisone in Men With Metastatic Castration-Sensitive Prostate Cancer or Non-Metastatic or Metastatic Castration-Resistant Prostate Cancer
Brief Title: Study of Relugolix in Men With Metastatic Castration-Sensitive Prostate Cancer or Non-Metastatic or Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MVT-601-049
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer; Metastatic Castration-Sensitive Prostate Cancer; Non-Metastatic Castration-Resistant Prostate Cancer
Keywords: mCRPC; mCSPC; Relugolix; Abiraterone; Prednisone; Leuprolide acetate; nmCRPC; Apalutamide; Docetaxel; Degarelix; Methylprednisolone
MeSH Terms: interventions — relugolix; abiraterone; Abiraterone Acetate; Prednisone; Methylprednisolone; apalutamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1: Relugolix plus Abiraterone plus a Corticosteroid (Experimental): Participants will receive relugolix in combination with abiraterone plus a corticosteroid for 12 weeks during the study treatment period.
  Interventions: Drug: Relugolix; Drug: Abiraterone; Drug: Prednisone; Drug: Methylprednisolone
- Part 2: Relugolix plus Apalutamide (Experimental): Participants will receive relugolix in combination with apalutamide for 12 weeks during the study treatment period.
  Interventions: Drug: Relugolix; Drug: Apalutamide
- Part 3: Relugolix plus Docetaxel with or without Prednisone (Experimental): Participants will receive relugolix in combination with docetaxel with or without prednisone for 12 weeks during the study treatment period.
  Interventions: Drug: Relugolix; Drug: Prednisone; Drug: Docetaxel

INTERVENTIONS:
Drug: Relugolix — (Part 1 and Part 3) Relugolix will be administered orally as a single 360-milligram (mg) loading dose of 3 x 120-mg tablets, followed by a 120-mg dose (1 x 120-mg tablets), taken once daily at approximately the same time each day.
  (Part 2) Relugolix will be administered orally as a single 360-milligram (mg) loading dose of 3 x 120-mg tablets, followed by a 240-mg dose (2 x 120-mg tablets), taken once daily at approximately the same time each day.
  Other Names: MVT-601; TAK-385; T-1331285; RVT-601; Orgovyx
Drug: Abiraterone — Abiraterone acetate (1000 mg [2 x 500-mg tablets]) or fine-particle abiraterone acetate (500 mg [4 x 125-mg tablets]) will be administered orally once daily.
  Other Names: Zytiga; Yonsa
  Arms: Part 1: Relugolix plus Abiraterone plus a Corticosteroid
Drug: Prednisone — (Part 1 only) For participants with mCSPC, a 5-mg dose of prednisone will be administered orally once daily, and for participants with mCRPC, a 5-mg dose of prednisone will be administered orally twice daily.
  (Part 3 only) Prednisone 5 mg can be administered orally twice daily but is not required.
  Arms: Part 1: Relugolix plus Abiraterone plus a Corticosteroid; Part 3: Relugolix plus Docetaxel with or without Prednisone
Drug: Methylprednisolone — For participants with mCRPC taking fine-particle abiraterone acetate, methylprednisolone 4 mg will be administered orally twice daily.
  Other Names: Medrol
  Arms: Part 1: Relugolix plus Abiraterone plus a Corticosteroid
Drug: Apalutamide — Apalutamide 240 mg (4 x 60-mg tablets) will be administered orally once daily.
  Other Names: Erleada
  Arms: Part 2: Relugolix plus Apalutamide
Drug: Docetaxel — Docetaxel 75 mg/m2 dose will be administered every 3 weeks as a 1-hour intravenous infusion.
  Other Names: Docefrez; Taxotere
  Arms: Part 3: Relugolix plus Docetaxel with or without Prednisone

SUMMARY:
This study is being conducted to assess the safety and tolerability of relugolix with other agents approved for use in combination with androgen deprivation therapy (ADT) for a 12-week treatment period and an additional 40-week safety extension period in men with prostate cancer, either metastatic castration-sensitive prostate cancer (mCSPC) or non-metastatic or metastatic castration-resistant prostate cancer (nmCRPC or mCRPC).

DETAILED DESCRIPTION:
This is a three-part, open-label, parallel-cohort study to assess the safety and tolerability of relugolix as the ADT component in combination treatment with abiraterone acetate plus a corticosteroid in patients with mCSPC or mCRPC (Part 1), apalutamide in patients with mCSPC or nmCRPC (Part 2), or docetaxel with or without prednisone in patients with mCSPC or mCRPC (Part 3).

The study will consist of a 45-day screening period followed by a 12-week treatment period with one of the three combination treatments (Parts 1, 2, or 3). All participants are required to be currently or previously treated with a GnRH receptor antagonist (analog), leuprolide acetate or triptorelin, or a GnRH receptor antagonist, degarelix or relugolix, in combination with either abiraterone plus prednisone (Part 1), apalutamide (Part 2), or docetaxel (Part 3). The study consists of a 12-week primary study treatment period in which safety and tolerability, including assessment of vital sign measurements, ECGs, clinical laboratory tests and reporting of adverse events every 2 to 4 weeks, followed by a 40-week safety extension treatment period during which adverse events and changes to concomitant medications will be reported. The total treatment duration is 52 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. A previous diagnosis of adenocarcinoma of the prostate confirmed by histologic or cytologic evidence and with a documented medical history of either:

   * mCSPC (Parts 1, 2, and 3) defined as having at least two of three risk factors at the baseline (Day 1) visit:

     * Total Gleason score of ≥ 6; and
     * Presence of ≥ 2 metastatic lesions on bone scan; OR
     * Radiologic evidence of measurable visceral metastases with exception of hepatic metastases.
   * nmCRPC (Part 2 only) defined as disease progression despite maintaining castration levels of testosterone with androgen deprivation therapy (ADT), as evidenced by an increase in consecutive prostate-specific antigen (PSA) concentrations (2 measurements, at least one week apart).
   * mCRPC (Parts 1 and 3) defined as disease progression despite maintaining castration levels of testosterone with ADT:

     * An increase in consecutive PSA (2 measurements at least 1 week apart); or
     * Worsening clinical symptoms; or
     * Radiologic evidence demonstrating enlarged metastatic lesions or the development of new metastases.
2. Initiating treatment or currently receiving treatment of leuprolide acetate (3-, 4-, or 6-month injections [intramuscular Lupron or subcutaneous Eligard]) or another GnRH receptor agonist (triptorelin) or a GnRH receptor antagonist (degarelix or relugolix [maximum duration of 3 months]) in combination with:

   * Part 1: abiraterone acetate 1000 mg or fine-particle abiraterone acetate 500 mg once daily plus prednisone 5 mg once daily for participants with mCSPC or twice daily for participants with mCRPC or methylprednisolone 4 mg once daily and in whom abiraterone has been well tolerated (that is, without evidence of hepatotoxicity requiring dose adjustment for abiraterone).
   * Part 2: apalutamide 240 mg once daily and in whom apalutamide has been well tolerated (that is, without a fracture, fall, or seizure episode or need to dose adjust due to any adverse events).
   * Part 3: docetaxel 75 mg/m2 and in whom docetaxel has been well tolerated (that is, no evidence of hypersensitivity reaction, febrile neutropenia or neutrophils < 500 cells/mm3 for more than 1 week, severe or cumulative cutaneous reactions, or moderate neurosensory signs and/or symptoms despite dose reduction). Note: Patients receiving treatment with another agent in addition to docetaxel, such as a steroid synthesis inhibitor or androgen receptor antagonist, may be enrolled.

Key Exclusion Criteria:

A patient will not be eligible for inclusion in the study if any of the following criteria apply:

1. A medical history of brain or hepatic metastases based on radiologic evidence or a medical history of surgical castration;
2. Received combination treatment with a GnRH analog or GnRH receptor antagonist with either abiraterone acetate plus a corticosteroid (Part 1) or apalutamide (Part 2) in patients with mCSPC (Part 1 and Part 2) or nmCRPC (Part 2) for a total duration > 24 months or in patients with mCRPC (Part 1) for a total duration > 6 months;
3. Is scheduled or anticipates being scheduled for major surgery during the study treatment period;
4. A current diagnosis of a malignancy other than prostate cancer, with the exception of any of the following:

   * Adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, or carcinoma in situ of any type;
   * Adequately treated Stage I cancer that is currently in remission and has been in remission for ≥ 2 years;
   * Any other cancer from which the patient has been disease-free for ≥ 3 years;
5. Abnormal clinical laboratory test value(s) at the screening visit or prior to the baseline (Day 1) visit including:

   * Serum creatinine > 2.0 mg/dL;
   * Platelets < 100 × 103/μL;
   * Hemoglobin < 10.0 g/dL;
   * Leukocytes (WBC) < 3 × 103/μL;
   * Absolute neutrophil count < 1.5 × 103/μL;
   * Hemoglobin A1c (HbA1c) > 8%; Note (Part 3 only): Transfusions and/or administration of growth factors are permitted as indicated for the clinical management of docetaxel-related hematologic effects and in accordance with the investigator's judgement.
6. Known hepatic disease, including alcoholic liver disease or viral hepatitis such as hepatitis A (hepatitis A virus IgM positive), chronic hepatitis B (HbsAg positive), or chronic hepatitis C (HCV antibody positive, confirmed by HCV RNA) or clinical signs of hepatic disease such as jaundice;
7. A medical history within 6 months prior to the screening visit or a current diagnosis of any of the following:

   * Myocardial infarction;
   * Unstable angina;
   * Unstable symptomatic ischemic heart disease;
   * Congestive heart failure classified as NYHA class III or IV heart failure;
   * Thromboembolic event(s) (eg, deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular event[s]);
   * Any other significant cardiac condition (eg, pericardial effusion, restrictive cardiomyopathy, severe untreated valvular stenosis, or severe congenital heart disease);
8. An abnormal ECG;
9. Uncontrolled hypertension;
10. Hypotension;
11. Bradycardia;
12. Positive HIV;
13. Medical history of a bleeding disorder or current clinical evidence of gastrointestinal bleeding or active bleeding from another anatomical location;
14. A medical history within 1 year of the screening visit of drug or alcohol abuse disorder according to Diagnostic and Statistical Manual of Mental Disorders V;
15. Received an investigational drug within 28 days or 5 half-lives, whichever is longer, prior to the baseline (Day 1) visit;
16. Prior use of any prohibited medication(s) and restrictive medication(s) without the appropriate washout period or use of a prohibited medication during the study treatment period is planned;
17. A contraindication or known history of hypersensitivity to any of the study treatments or components thereof, or has a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates study participation;
18. Any other medical or psychiatric condition that, in the opinion of the investigator, would interfere with accomplishing the study objectives or the patient completing the study;
19. Is a study site employee or is a primary family member (spouse, parent, child, or sibling) of a site employee involved in the conduct of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Baseline through Week 13
  Parts 1, 2, and 3

SECONDARY OUTCOMES:
Mean Testosterone Serum Concentrations at Baseline (Day 1), Week 5, and Week 13 | Baseline (Day 1), Week 5, and Week 13
  Parts 1 and 2
Number and Proportion of Participants with Testosterone Concentrations ≥ 50 ng/dL at Baseline (Day 1), Week 5, and Week 13 | Baseline (Day 1), Week 5, and Week 13
  Parts 1 and 2
Relugolix Trough Concentrations at Baseline (Day 1), Week 3, Week 5, Week 9, and Week 13 | Baseline (Day 1), Week 3, Week 5, Week 9, and Week 13
  Part 2
Apalutamide and N-desmethyl Apalutamide Trough Concentrations at Baseline (Day 1), Week 3, Week 5, Week 9, and Week 13 | Baseline (Day 1), Week 3, Week 5, Week 9, and Week 13
  Part 2
Mean Testosterone Serum Concentrations at Baseline (Day 1), Mid-Treatment, and Week 13 | Baseline (Day 1), Mid-Treatment, and Week 13
  Part 3
Number and Proportion of Participants with Testosterone Concentrations ≥ 50 ng/dL at Baseline (Day 1), Mid-Treatment (Treatment Cycle that Most Closely Corresponds to Week 7 of the Primary Study Treatment Period), and Week 13 | Baseline (Day 1), Mid-Treatment (Treatment Cycle that Most Closely Corresponds to Week 7 of the Primary Study Treatment Period), and Week 13
  Part 3
Relugolix Concentrations at Baseline (Day 1), In-Cycle, Mid-Treatment, and Week 13 in Each Infusion Cycle for Docetaxel | Baseline (Day 1), In-Cycle, Mid-Treatment, and Week 13 in Each Infusion Cycle for Docetaxel
  Part 3
Docetaxel Concentrations at Baseline (Day 1), In-Cycle, Mid-Treatment, and Week 13 in Each Infusion Cycle for Docetaxel | Baseline (Day 1), In-Cycle, Mid-Treatment, and Week 13 in Each Infusion Cycle for Docetaxel
  Part 3
Incidence of Adverse Events | Up to 52 weeks
  Parts 1, 2, and 3

CONTACTS AND LOCATIONS:
Overall Officials: Mike Ufer, Study Director — Sumitomo Pharma America, Inc.
Locations (16):
- United States (16):
  - Urological Associates of Southern Arizona, P.C., Tucson, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - Colorodo Clinical Research, Lakewood, Colorado
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - New Jersey Urology, Saddle Brook, New Jersey
  - Clinical Research Alliance, Inc., Westbury, New York
  - Alliance Urology, Greensboro, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Helios Clinical Research, LLC., Middleburg Heights, Ohio
  - Center for Advanced Urology, LLP d/b/a: MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Urology San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De La Cerda J, Belkoff L, Courtney KD, Diamond E, D'Olimpio J, Dunshee C, Gervasi L, Goodman M, Mittal K, Morris D, Sieber P, Tutrone R, Ryan M, Zhong Y, Ufer M, Shore N. Safety and Tolerability of Relugolix in Combination with Abiraterone or Apalutamide for Treatment of Patients with Advanced Prostate Cancer: Data from a 52-Week Clinical Trial. Target Oncol. 2025 May;20(3):503-517. doi: 10.1007/s11523-025-01139-3. Epub 2025 Apr 4. PMID 40180682
- [Derived] De La Cerda J, Dunshee C, Gervasi L, Sieber P, Belkoff L, Tutrone R, Lu S, Gatoulis SC, Brown B, Migoya E, Shore N. A Phase I Clinical Trial Evaluating the Safety and Dosing of Relugolix with Novel Hormonal Therapy for the Treatment of Advanced Prostate Cancer. Target Oncol. 2023 May;18(3):383-390. doi: 10.1007/s11523-023-00967-5. Epub 2023 Apr 15. PMID 37060432